CLINICAL TRIAL: NCT00957320
Title: A Phase I Study of Sirolimus With PEG-Asparaginase in Multiple Recurrent or Refractory Childhood Acute Lymphoblastic Leukemia
Brief Title: Study of Sirolimus With PEG-Asparaginase in Acute Lymphoblastic Leukemia (ALL)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no patients enrolled, decided not to pursue study
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Frank Keller, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00015324; Sirolimus (Other: Other)
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: leukemia; cancer; oncology; sirolimus; ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Neoplasms | interventions — Sirolimus; pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Subjects will receive PEG-asparaginase at a fixed weekly dose, as per published reports in relapsed childhood ALL. The dose of sirolimus will be dose escalated following standard phase 1 statistical methods.
  For patients with active CNS leukemia, intrathecal methotrexate, hydrocortisone and cytarabine (triple IT) will be administered weekly, with leucovorin rescue at the treating physician's discretion.
  Interventions: Drug: Sirolimus; Drug: PEG-asparaginase

INTERVENTIONS:
Drug: Sirolimus — Sirolimus daily po days 1 through 28, Dose level 0: 0.25 mg/m2 po daily Dose level 1: 0.5 mg/m2 po daily Dose level 2: 1 mg/m2 po daily Dose level 3 1.5 mg/m2 po daily Dose level 4 2 mg/m2 po daily
Drug: PEG-asparaginase — Subjects will receive PEG-asparaginase at a fixed weekly dose, as per published reports in relapsed childhood ALL.

SUMMARY:
The goal of this study is to find a safe dose of sirolimus that can be used with a standard dose of L-asparaginase. To find the safe dose, the investigators will give the first patient a very small dose of sirolimus (smaller than the dose used in organ transplant children) and the standard dose of L-asparaginase. The investigators will then look for side effects. If side effects develop, the investigators will decrease the dose of sirolimus. If they do not, the investigators will increase the dose of sirolimus in the next patient on the study. The investigators will continue this method until fewer than one-third of patients have a side effect that would require stopping the drug or changing the dose.

The investigators plan to enroll up to 15 children with relapsed ALL. The enrolled patients must have recovered from other treatment before starting this study. Also, they cannot have severe side effects from their earlier therapy that will possibly make these drugs less safe.

The investigators will collect information on whether these drugs help to cure the ALL, but the purpose will be to find a dose of sirolimus that does not cause too many side effects when combined with L-asparaginase. This will be explained to the families and they will sign a written consent. The patients will provide either verbal or written assent when appropriate.

DETAILED DESCRIPTION:
Multiple relapsed acute lymphoblastic leukemia (ALL) has a very poor cure rate, and there is no standard of care for treatment of these patients. Therefore, we want to combine two chemotherapy drugs to see if they are safe and will help treat these patients. The first agent, L-asparaginase, is used in most patients during their initial treatment for ALL. The second agent, sirolimus, causes death in human leukemia cells in the laboratory. Sirolimus is also used in children who have received kidney or heart transplants to prevent organ rejection. Therefore, the safety and side effects are well known in children.

There are many steps that allow cancer cells to grow in humans. L-asparaginase and sirolimus block two different steps in cell growth. Because of this, we anticipate that these two drugs will work together to lead to more cancer cell death.

The first part of the study will last 1 month for each patient. If the patients have a good response to these two drugs, they will be allowed to continue these drugs for up to 12 months. They will continue on the dose of sirolimus that they received during the first month for the remaining time on the study.

We will also look at the way leukemia cells are responding to these medications in the laboratory. We will not draw any blood or bone marrow samples from the patient unless they already need the procedure done for other tests. The amount of extra blood or bone marrow drawn will not cause the patients any harm. As we do not know what these laboratory tests mean, we will not tell the patients the results during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Less than 21 years old.
2. Acute lymphoblastic leukemia.
3. Second or greater bone marrow relapse or 1st relapse and refractory to at least 2 Attempts at re-induction.
4. Life expectancy of at least 8 weeks.
5. Fully recovered from the acute toxic effects of all prior therapy.
6. Appropriate organ function.

Exclusion Criteria:

1. Patients with a documented history of ≥ grade 3 local or systemic reactions to PEG-asparaginase.
2. Patients with a documented history of anti-E. coli asparaginase antibodies.
3. Patients with a history of ≥ grade 3 pancreatitis.
4. Patients with an active and uncontrolled infection.
5. Patients s/p allogeneic bone marrow transplantation, who are still on immunosuppressants.
6. Pregnant or lactating females. Women of childbearing age will agree to use contraception during the protocol.
7. Patients currently receiving other investigational agents, medications, or supplements with a known anti-leukemic effect.
8. Other concomitant medications that may alter the metabolism of Sirolimus (See section 7.2).
9. Patients who, in the opinion of the investigator, will not be able to comply with safety monitoring requirements of the study.
10. Patients with a history of a documented thrombus from previous asparaginase therapy.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To estimate the maximum tolerated dose (MTD) of sirolimus in children with refractory or recurrent acute lymphoblastic leukemia (ALL) who are concurrently receiving PEG-asparaginase. | end of study
To determine the dose limiting toxicities of sirolimus in combination with PEG-asparaginase in this Phase I Study. | end of study

SECONDARY OUTCOMES:
To use phospho-flow to measure the degree of phosphorylation of signaling pathway proteins in response to specific stimulating events in bone marrow derived leukemia cells obtained at the time of study entry and at day 15 and 29. | end of study
To correlate the signal pathway phosphorylation to clinical response to the chemotherapy regimen used in this study. | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Frank Keller, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States